CLINICAL TRIAL: NCT05028972
Title: Implementing HearVA (I-HearVA)
Brief Title: Hearing Impairment, Strategies and Outcomes in VA Emergency Departments
Acronym: HearVA-ED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 17-068-1; HX002421 (Other Grant/Funding Number: VA HSR&D)
Record Dates: First submitted 2021-08-24; First posted 2021-08-31 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Hearing Loss; Emergency Service; Hospital Readmission
Keywords: Hearing loss; Emergency service; ED Revisit; Communication
MeSH Terms: conditions — Hearing Loss; Communication

STUDY DESIGN:
Intervention Model Description: Consenting participants will be randomly assigned to the control or intervention arm of the study. Participants in the intervention arm will receive PockeTalkers (personal amplifiers) for the duration of their time in the emergency department. Participants in the control group will not receive personal amplifiers during their time in the emergency department, but will receive one upon discharge from the emergency department. In later stages, there will be no control group and all participants will receive a personal amplifier during their time in the emergency department.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention: Personal Amplifier (Experimental): Consenting participants will be randomly assigned to the intervention group while receiving care in the emergency department
  Interventions: Other: Personal Amplifier
- Control: No Personal Amplifier (Other): Consenting participants will be randomly assigned to the control group while receiving care in the emergency department
  Interventions: Other: No Personal Amplifier

INTERVENTIONS:
Other: Personal Amplifier — The intervention group will receive personal amplifiers (PockeTalkers) while they receive care in the ED
  Other Names: Pocketalker
  Arms: Intervention: Personal Amplifier
Other: No Personal Amplifier — The control group will not receive personal amplifiers while they receive care in the ED
  Arms: Control: No Personal Amplifier

SUMMARY:
HearVA involves six VA facility emergency departments (ED) over a 3-year intervention period. The first part of this study will test whether providing personal amplifiers to Veteran ED patients who self-report hearing difficulty is acceptable to these patients, can improve their hearing, enhance understanding of discharge instructions, and can reduce the risk of coming back to the ED in a short period of time (3 days and 30 days). The second part of the study will then identify whether ED staff can implement this program and achieve similar results. The second part will give ED staff increasing levels of responsibility for screening Veterans for hearing difficulty and providing personal amplifiers when such difficulty is detected.

DETAILED DESCRIPTION:
HearVA is a randomized controlled trial to explore the utility and outcomes of providing point-of-care access to hearing-impaired Veterans, comparing an offer of personal amplifiers versus control in an environment where the clinical stakes are high. It addresses a knowledge gap about the utility of providing such hearing assistance during clinical encounters. The study measures whether providing personal amplifiers is acceptable to older patients, can improve hearing, enhance understanding of discharge instructions, and improve care transitions at discharge. If such a strategy is beneficial, this simple low-tech approach has great potential for implementation and wide dissemination. HearVA-ED has two phases - the first, which has been completed, established the feasibility and acceptability of research and procedures in the ED environment through a pilot efficacy study and the second phase will be to complete a larger more definitive efficacy study and a detailed implementation study resulting in a strategic approach that can be widely disseminated across all VA emergency departments throughout the United States. This second phase will use a mixed-methods, hybrid effectiveness-implementation design to implement and evaluate the hearing assistance intervention in six VA Emergency Department Sites (in different facilities across the country). Implementation will occur in four stages with variation in the starting sequence at each site: The first group of two VA emergency departments will initiate implementation with an efficacy trial; second group of two sites will initiate implementation with delivery and support of personal amplifiers after screening and randomization by a research assistant (Stage 1); the third group of two sites will initiate implementation with the entire implementation (Stage 2) and the presence of a research assistant to conduct discharge interviews; and all sites will progress from this sequence to Stage 3 - Sustainability - which is the full implementation without research assistant presence.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Emergency severity index criterion of 3 (medium), 4, or 5 (low acuity)
* Hearing Handicap Inventory-Screen greater than or equal to 10 or positive answer to a single-item screening question
* Capacity to consent to participate in research

Exclusion Criteria:

* Inability to consent to participate in research
* Emergency severity index criterion of 1-2 (high acuity)
* Hearing Handicap Inventory-Screen less than 10 and negative answer to single item screening question
* Inability to speak English
* Using cochlear implants

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Estimated)
Dates: Start 2021-12-08 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
ED 3-day Readmissions | 3-5 days after initial ED stay
  The Investigators will determine whether patients have had an ED revisit within three days through CPRS review as well as a brief follow-up phone call 3-5 days after ED discharge

SECONDARY OUTCOMES:
ED 30-day Readmissions | 30-35 days after initial ED stay
  The Investigators will determine whether patients have had an ED revisit within 30 days through CPRS review as well as a brief follow-up phone call 30-35 days after ED discharge
Patient-Rated Quality of Hearing, Understanding, and Communication With Providers During ED Stay | Duration of ED stay, average of 1 day
  Participants will self-rate their quality of hearing, understanding, and communication using a six item questionnaire. Scored on a 10-point Likert scale (1 = do not agree at all; 10 = completely agree) the questions will be: When I talked to the doctors and nurses today ... (1) their voices were very clear; (2) I was able to hear the sounds that I wanted to hear; (3) noises did not cause a problem for my hearing; and (4) listening did not make me tired. Two additional statements will explicitly capture understanding: (5) I was able to understand what they said; and (6) I was able to understand without making an effort. Higher scores will indicate better communication and understanding with providers.
Patient-Rated Quality of Post-Discharge Care | At time of discharge from ED, average 1 day
  Patient-rated quality of post-discharge care using a three-item subset of the Care Transition Measure (CTM). The questions are scored on a 1-4 scale (1= strongly disagree; 4 = strongly agree): (1) The ED staff considered my preferences and those of my family or caregiver in deciding what my healthcare needs were for discharge; (2) Leaving the ED, I have a good understanding of the things I am responsible for in managing my health; (3) Leaving the ED, I clearly understand the purpose for each of my medications. Higher scores will indicate better discharge preparation.
Self-Reported Understanding of Discharge Instructions | 3-5 days after initial ED stay
  Investigators will gauge self-reported understanding of discharge instructions using semi-structured interview data compared to documented discharge data.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Chodosh, MD MSHS, Principal Investigator — VA NY Harbor Healthcare System, New York, NY
Locations (6):
- United States (6):
  - Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado
  - VA NY Harbor Healthcare System, New York, NY, New York, New York
  - Syracuse VA Medical Center, Syracuse, NY, Syracuse, New York
  - James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No